CLINICAL TRIAL: NCT01575340
Title: Markers of the Inflammatory Response (IL-1β, IL-10, IL-17A and TNF-α) in Patients With Colorectal Cancer in Chemotherapy Supplemented With Fish Oil
Brief Title: Study to Assess the Effect of Consumption of Fish Oil Encapsulated on Inflammatory Markers in Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Collaborators: Fundação de Amparo à Pesquisa e a Inovação do Estado de Santa Catarina (Unknown); Centro de Pesquisas Oncológicas de Florianópolis (Unknown)
Responsible Party: Principal Investigator, Erasmo Benicio Santos de Moraes Trindade, Clinical Professor, Universidade Federal de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20.179/2010-0
Record Dates: First submitted 2011-10-05; First posted 2012-04-11 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Cancer; Inflammation
Keywords: inflammatory markers; colorectal cancer; cytokines; fish oil
MeSH Terms: conditions — Colorectal Neoplasms; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fish oil encapsuled (Experimental): will receive the supplementation of 2 g / day of fish oil encapsulated for 9 weeks
  Interventions: Dietary Supplement: fish oil encapsuled
- without supplementation (No Intervention): not will receive supplementation or encapsulated fish oil or placebo

INTERVENTIONS:
Dietary Supplement: fish oil encapsuled — 2 g/d (4 capsules of 500 mg)for 9 weeks
  Other Names: omega-3 encapsuled
  Arms: fish oil encapsuled

SUMMARY:
The purpose of this study is to evaluate whether supplementation 2g/day encapsulated fish oil modifies inflammatory markers in individuals with colorectal cancer in chemotherapy

DETAILED DESCRIPTION:
The study will recruit patients with newly diagnosed colorectal cancer and that has not yet undergone any chemotherapy treatment. Individuals that meet the inclusion criteria are randomized by means of a computer program on two study groups: 1) supplemented Experimental: receive 2g/day supplementation encapsulated fish oil for 9 weeks. 2) No intervention - control: not receive supplementation of fish oil or placebo. Will be assessed the effects of supplementation on the standard profile of cytokine production, nutritional status, and proportion of incorporation of these fatty acids in blood cells (mononuclear and red blood cells).

Blood samples are collected before the start of first chemotherapy and nine weeks later. Supplementation in the experimental group also will start on the first day of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years
* Histopathological diagnosis of colorectal cancer
* Beginning of chemotherapy in the target institution
* Agree to participate in the study [signature of IC]

Exclusion Criteria:

* Age <19 years
* Being in palliative care
* Inability to oral intake
* Allergic to the fish and fish products
* Owning with hyperlipidemia requiring drug treatment
* Consumption prior to the study of fish oil or supplements containing omega-3 PUFA
* Being in medical treatment with some nonsteroidal anti-inflammatory
* Have some kind of infection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-07; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
change in inflammatory markers | two months
  will be evaluated cytokines IL-1 beta, IL-10, IL-17A and TNF alpha, and acute phase proteins CRP and Albumin, in baseline that corresponds to the day that the patient will begin chemotherapy and the final moment, which corresponds to 9 weeks counting from the baseline in both groups (supplemented and non-supplemented)

SECONDARY OUTCOMES:
change in body composition | two months
  will estimate the percentage of body fat in each patient through the use of skinfold thickness at baseline and end to study in both groups
change in nutritional status | two months
  will be measured anthropometric measures: weight and height (baseline and end of study) for the classification of nutritional status according to BMI
Changes in plasma lipid profile | two months
  will evaluate the proportion of incorporation of omega-3 fatty acids in plasma
assessing the risk of inflammatory and nutritional complications | two months
  Will be calculated the ratio PCR / albumin, as proposed by Correa et al., 2002, using the cutoff points proposed by the same author for the classification of high, medium, decreased or no risk

CONTACTS AND LOCATIONS:
Overall Officials: Michel C Mocellin, Master's, Principal Investigator — Universidade Federal de Santa Catarina
Locations (1):
- Centro de Pesquisas Oncológicas - CEPON, Florianópolis, Santa Catatina, Brazil